CLINICAL TRIAL: NCT06952244
Title: Investigation of Clinical and Functional Characteristics of Endocrinology Patients During Hospitalization
Brief Title: Functional Status in Hospitalized Endocrine Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Principal Investigator, Uşak University
Other Study IDs: 561-561-10
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Endocrine Diseases; Hospitalized
Keywords: endocrine diseases; functional assessment; clinical assesment; Hospitalization; Individuals with endocrine disorders
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized in the endocrinology ward: patients in the endocrinology service will be accepted to Uşak training and research hospital with a doctor's diagnosis. General physical, functional and psychosocial and blood values evaluations will be made.

SUMMARY:
The aim of this observational study was to examine the clinical and functional characteristics of patients hospitalized in the endocrinology department of a university hospital. In line with this purpose, the following research questions were given.

What are the respiratory functions and respiratory rates of patients hospitalized in the endocrinology department? What are the muscle strengths of patients hospitalized in the endocrinology department? What is the general health status of patients hospitalized in the endocrinology department? What is the quality of life of patients hospitalized in the endocrinology department? What is the fatigue status of patients hospitalized in the endocrinology department? What is the level of independence of patients hospitalized in daily living activities of patients hospitalized in the endocrinology department? What are the routine blood values of patients hospitalized in the endocrinology department? What is the sleep quality of patients hospitalized in the endocrinology department? What are the physical activity levels of patients hospitalized in the endocrinology department? What is the balance status of patients hospitalized in the endocrinology department? What is the neuropathic pain status of patients hospitalized in the endocrinology department? The patients hospitalized in the Endocrinology Department of Uşak Education and Research Hospital constitute the sample of the study. Clinical and functional evaluations will be made from the participants during their hospital stay. In this context, respiration, muscle strength, general pain assessment, life expectancy, fatigue, independence levels, sleep quality, routine blood values, physical activity levels, balance status and neuropathic status evaluation will be made.

DETAILED DESCRIPTION:
The endocrine system is a system responsible for the production of hormones that regulate vital functions such as metabolism, growth, reproduction and energy balance. Endocrine diseases can seriously affect the general health status, functional capacity and quality of life of individuals by causing disruptions in these functions. Endocrine patients usually require hospitalization due to chronic symptoms caused by metabolic and hormonal imbalances. During this process, negative changes may occur in many clinical, physical and functional characteristics.

Clinical Features: Parameters such as routine blood values, respiratory functions and muscle strength play a critical role in monitoring the general health status of patients.

Functional Features: Factors such as independence in daily living activities, balance, physical activity level and sleep quality are important elements that should be evaluated during the hospitalization period of patients.

Main Problems Encountered by Endocrinology Patients Metabolic Problems: Conditions such as hyperglycemia, hypoglycemia, electrolyte imbalances and insulin resistance are frequently seen.

Loss of Muscle and Functional Capacity: Endocrine diseases can negatively affect muscle strength and limit the independence and daily living activities of individuals.

Sleep and Fatigue Problems: Hormonal imbalances can reduce quality of life by affecting sleep quality and energy levels.

Balance and Coordination Difficulties: Complications such as diabetic neuropathy can affect neuromuscular functions and lead to balance problems.

Psychosocial Effects: Psychological effects such as chronic fatigue, depression, and decreased quality of life have been widely reported. This study aims to comprehensively evaluate the conditions of endocrinology patients during their hospitalization and understand the relationship between both clinical and functional characteristics. Such an approach provides basic data for better management of patients, development of treatment protocols, and improvement of hospitalization processes.

Focus Points of the Study Sociodemographic Characteristics Examination: Understanding the effects of factors such as age, gender, and education level on clinical and functional outcomes.

Analysis of Clinical Parameters: Evaluating the role of biophysical measurements such as routine blood values and respiratory functions in the disease process.

Functional Capacity Assessment: Determining the effects of muscle strength, balance, and physical activity levels on daily life.

Measuring Quality of Life: To investigate how health-related quality of life is affected by factors such as sleep quality and fatigue.

Research on endocrine diseases shows that these patients often face long hospitalization periods, high risk of complications, and reduced quality of life. Measurements such as muscle strength, respiratory function, and balance are used to estimate both the health status of individuals and the recovery process. Quality of life is affected not only by physical health but also by psychosocial and environmental factors. The findings of this study can be used to determine the difficulties experienced by endocrine patients during the hospitalization process and areas for improvement during this process. It can also guide the development of individualized treatment and rehabilitation programs. Based on this, the aim of the study was to examine the clinical and functional characteristics of patients hospitalized in the endocrinology department of a university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-64
* Being a volunteer
* Being hospitalized in the endocrinology ward.

Exclusion Criteria:

* Patients who have any obstacles to participating in surveys and measurements,
* Patients with missing data for any reason, and patients who are not accepted to the endocrinology service

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample of the study consists of patients aged between 18-64 years who are hospitalized in the Endocrinology Department of Uşak Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of respiratory functions | At the time of enrollment
  Respiratory rate: Respiratory rate provides important information in the diagnosis of respiratory problems and in the evaluation of the general health status of the individual. The number of breaths the individual takes in a minute (how many times the chest rises) will be counted. During the evaluation, the hands will be placed on the patient's chest and the movements in the chest wall will be felt and the counts made during rest, inspiration and expiration will be evaluated.
Chest circumference measurement | At the time of enrollment
  Chest circumference measurement: Respiratory function is an important parameter for monitoring and evaluating respiratory functions. The measurement will be taken at the level of the fourth rib, where the lower end of the scapula passes, while standing with the arms abducted. The measurement will be made twice during rest, inspiration and expiration. Thus, chest mobility will also be evaluated.
Assessment of muscle strength | At the time of enrollment
  Manual Muscle Testing: Manual muscle testing is used to assess the muscle strength of individuals and identify possible weaknesses or imbalances. The strength of large muscle groups such as quadriceps femoris and biceps brachii is essential for individuals to carry out their daily activities. Weakness in these muscles can negatively affect a person's independence and quality of life. In our study, muscle strength will be assessed with a score between 0 and 5 (0: no muscle contraction is felt, 5: full movement of the segment against gravity and with maximum resistance).
Pain assessment | At the time of enrollment
  Pain assessment will be done with Visual Analog Scale (VAS). VAS includes a scale with a starting and ending point on a line to evaluate a specific feature. Individuals evaluate the severity of their condition by placing a mark on this line. In this scale, 0 represents the absence of a specific feature or no sensation, and 10 represents the highest intensity of that feature. In our study, it was used to evaluate general health status.
Quality of life assessment | At the time of enrollment
  Short Form-36 Health Survey (SF-36) was developed by John E. Ware and colleagues (1992) to measure health-related quality of life. It consists of a total of 36 questions covering physical, psychological and social dimensions. Sub-dimensions: Physical Function, Social Function, Body Pain, General Health, Mental Health, Vitality, Physical Role and Emotional Role. Scores calculated for each subscale range from 0 to 100, where higher scores indicate better health status, functioning and quality of life.
Fatigue assessment | At the time of enrollment
  Functional Assessment of Chronic Illness Therapy (FACIT): FACIT is a scale developed to assess the level of fatigue that individuals experience, particularly due to chronic diseases. This scale, consisting of a total of 13 questions, measures the level of fatigue and energy experienced by individuals in the last week. Each item on the FACIT scale is scored between 0 and 4; responses range from "never" to "very often." The total score obtained ranges from 0 to 52, with higher scores indicating lower fatigue and better quality of life.
Assessing their independence in activities of daily living | At the time of enrollment
  Assessment of independence in daily living activitiesBarthel Index: It will be assessed with the Barthel Index. The Barthel index was developed by Florence I. Mahoney and Dorothy W. Barthel in 1965. It is used to assess the level of independence in daily living activities. Scoring: Scored between 0-100. Higher scores mean more independence. The areas of use of this index are rehabilitation, post-stroke independence assessment, neurological and geriatric patients. It is a short and easy-to-use index.
Routine Blood Values Examination | At the time of enrollment
  Routine blood tests consist of standard biochemistry, hemogram, and electrolyte tests that evaluate the general health status of the individual. This assessment was not developed by any specific author; it is standardized by medical guidelines and laboratory practices.
Evaluation of sleep quality | At the time of enrollment
  PSQI (Pittsburgh Sleep Quality Index): PSQI was developed by Daniel J. Buysse and colleagues (1989). It is used to evaluate sleep quality and sleep disorders. Sub-dimensions: Subjective Sleep Quality, Sleep Latency (Time to Fall Asleep), Sleep Duration, Sleep Efficiency, Sleep Disorders, Medication Use, Daytime Functioning. Scoring: Scored between 0-21; 5 and above indicates poor sleep quality.
The physical activity level | At the time of enrollment
  The physical activity level will be assessed. The International Physical Activity Questionnaire (IPAQ) was developed by the World Health Organization and an international consortium. It is a standard tool for assessing physical activity level. This questionnaire was developed by Craig et al. (2003). The scale has 3 categories. These are: Categories: Low Activity, Moderate Activity, High Activity. It is a questionnaire frequently used in studies related to sports sciences, public health and physical activity level.
Balance assessment | At the time of enrollment
  Balance assessment will be evaluated with the Berg Balance Scale. The Berg Balance Scale was developed by Katherine Berg and her colleagues in 1992. The Berg Balance Scale is a clinical assessment tool used to assess individuals' risk of falling, measure functional balance levels, and monitor the effectiveness of rehabilitation programs. Total Number of Items on the Scale: 14 items. Scoring: Each item is scored between 0 and 4 (0 = cannot perform the task, 4 = performs the task completely). Total Score Range: 0-56.
Neuropathy evaluation | At the time of enrollment
  Neuropathy assessment will be done with the Michigan Neuropathy Assessment Questionnaire. The Michigan Neuropathy Assessment Questionnaire was developed by William H. Herman and colleagues (1994). It is used to assess diabetic neuropathy. The questionnaire asks about the patient's neuropathy symptoms (tingling, numbness, pain in the feet, etc.). Clinical assessment findings such as tenderness in the feet, loss of reflexes, and thinning of the skin will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gursan, Dr., Principal Investigator — Uşak University
Locations (1):
- Uşak Education and Research Hospital, Uşak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to protect participant confidentiality and comply with the confidentiality commitment approved by the ethics committee, no sharing of individual-level data is planned. In addition, the ethics committee decision that approved the study covers data use with limited access only. Therefore, it may not be possible to share IPD data publicly.